CLINICAL TRIAL: NCT01570400
Title: Reduction of Social Phobia Symptoms With Combined Internet-Based Cognitive Bias Modification and Cognitive Behavioral Therapy
Brief Title: Treatment of Social Phobia With Combined Cognitive Bias Modification and iCBT
Acronym: SOFIE13a
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Per Carlbring, PhD, Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOFIE13a
Record Dates: First submitted 2012-03-29; First posted 2012-04-04 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Social Phobia
Keywords: social phobia; social anxiety; cognitive bias modification
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBM training program variant 1 + iCBT (Experimental): Cognitive bias modification training program variant 1 combined with iCBT
  Interventions: Behavioral: Internet-administered cognitive behavioral therapy (iCBT); Behavioral: Cognitive bias modification training program variant 1
- CBM training program variant 2 + iCBT (Experimental): Cognitive bias modification training program variant 2 combined with iCBT
  Interventions: Behavioral: Internet-administered cognitive behavioral therapy (iCBT); Behavioral: Cognitive bias modification training program variant 2

INTERVENTIONS:
Behavioral: Internet-administered cognitive behavioral therapy (iCBT) — Established form of internet-administered cognitive behavioral therapy. Controlled progress, self-help modules with psychoeducative texts, assignments and homework. Therapist assisted.
Behavioral: Cognitive bias modification training program variant 1 — Computerized, internet-based training program for implicit modification of cognitive bias of attention, variant 4. Participant is exposed to a pair of words or a pair of faces -- either neutral-negative, neutral-positive, or negative-positive -- for 500ms-1000ms, followed by a probe (< or >) in the previous position of ONE of these words or faces and is then asked to press the corresponding arrow button on a keyboard. A total of 96 word pairs and 96 face pairs are shown during a session. One third is neutral-negative, one third is neutral-positive, and one third is negative-positive. The probe always follows the more negative word or face.
  Duration: approx. 10 min. per session. Frequency: Once every day for 2 weeks.
  Arms: CBM training program variant 1 + iCBT
Behavioral: Cognitive bias modification training program variant 2 — Computerized, internet-based control training program, variant 2. Participant is exposed to a pair of words or a pair of faces -- either neutral-negative, neutral-positive, or negative-positive -- for 500ms-1000ms, followed by a probe (< or >) in the previous position of ONE of these words or faces and is then asked to press the corresponding arrow button on a keyboard. A total of 96 word pairs and 96 face pairs are shown during a session. One third is neutral-negative, one third is neutral-positive, and one third is negative-positive. The probe follows the more positive stimulus and the more negative stimulus with equal frequency.
  Duration: approx. 10 min. per session. Frequency: Once every day for 2 weeks.
  Arms: CBM training program variant 2 + iCBT

SUMMARY:
The purpose of this study is to determine whether an internet-based treatment program, consisting of combined cognitive bias modification and cognitive behavioral therapy, reduces symptoms of social phobia among a population diagnosed with this disorder.

DETAILED DESCRIPTION:
Previous studies have shown that individuals with social phobia have attention biases, often focusing on or avoiding aversive stimuli (such as judging facial expressions) and thereby reinforcing the bias. Computerized training programs have been developed to implicitly direct the users attention. In this study, such a program -- combined with an established, well-researched and proven effective form of internet-based cognitive behavioral therapy (iCBT) -- will be provided to 128 participants that meet the diagnostic criteria for social phobia, and the pre/post-measurements will be compared. Participants will be randomized to one of two groups, receiving one of two variants of the cognitive bias modification program (both receive iCBT).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided
* Diagnosed social phobia (according to DSM-IV criteria)
* Access to computer with internet connection

Exclusion Criteria:

* Severe depression (and/or suicidal behavior)
* Suffer from other severe psychiatric condition (e.g. psychosis)
* Non-stable use of medication (3 months stable dosage)
* Undergoing other, parallel psychological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Liebowitz Social Anxiety Scale Self-Rated (LSAS-SR) | 24 hours
  The Liebowitz Social Anxiety Scale (LSAS) is a questionnaire by psychiatrist and researcher, Michael Liebowitz, whose objective is to assess the range of social interaction and performance situations which patients with social anxiety disorder may fear. It is commonly used to study outcomes in clinical trials. The scale features 24 items, 13 relating to performance anxiety and 11 concerning social situations. It is not intended for use as a self-reporting diagnosis.
Change from baseline in Liebowitz Social Anxiety Scale Self-Rated (LSAS-SR) | 11 weeks
  The Liebowitz Social Anxiety Scale (LSAS) is a questionnaire by psychiatrist and researcher, Michael Liebowitz, whose objective is to assess the range of social interaction and performance situations which patients with social anxiety disorder may fear. It is commonly used to study outcomes in clinical trials. The scale features 24 items, 13 relating to performance anxiety and 11 concerning social situations. It is not intended for use as a self-reporting diagnosis.
Change from baseline in Liebowitz Social Anxiety Scale Self-Rated (LSAS-SR) | 4 months
  The Liebowitz Social Anxiety Scale (LSAS) is a questionnaire by psychiatrist and researcher, Michael Liebowitz, whose objective is to assess the range of social interaction and performance situations which patients with social anxiety disorder may fear. It is commonly used to study outcomes in clinical trials. The scale features 24 items, 13 relating to performance anxiety and 11 concerning social situations. It is not intended for use as a self-reporting diagnosis.
Change from baseline in Liebowitz Social Anxiety Scale Self-Rated (LSAS-SR) | Two weeks into treatment
  The Liebowitz Social Anxiety Scale (LSAS) is a questionnaire by psychiatrist and researcher, Michael Liebowitz, whose objective is to assess the range of social interaction and performance situations which patients with social anxiety disorder may fear. It is commonly used to study outcomes in clinical trials. The scale features 24 items, 13 relating to performance anxiety and 11 concerning social situations. It is not intended for use as a self-reporting diagnosis.

SECONDARY OUTCOMES:
Change from baseline in Quality Of Life Inventory (QOLI) | 24 hours
  The QOLI assessment yields an overall score and a profile of problems and strengths in 16 areas of life such as love, work and play. The QOLI test is a measure of positive psychology and positive mental health.
Change from baseline in Quality Of Life Inventory (QOLI) | 11 weeks
  The QOLI assessment yields an overall score and a profile of problems and strengths in 16 areas of life such as love, work and play. The QOLI test is a measure of positive psychology and positive mental health.
Change from baseline in Quality Of Life Inventory (QOLI) | 4 months
  The QOLI assessment yields an overall score and a profile of problems and strengths in 16 areas of life such as love, work and play. The QOLI test is a measure of positive psychology and positive mental health.
Change from baseline in Quality Of Life Inventory (QOLI) | 2 weeks into treatment
  The QOLI assessment yields an overall score and a profile of problems and strengths in 16 areas of life such as love, work and play. The QOLI test is a measure of positive psychology and positive mental health.
Change from baseline in Social Phobia Scale + Social Interaction Anxiety Scale | 24 hours
  Self-rated measurements of social anxiety/phobia.
Change from baseline in Social Phobia Scale + Social Interaction Anxiety Scale | 11 weeks
  Self-rated measurements of social anxiety/phobia.
Change from baseline in Social Phobia Scale + Social Interaction Anxiety Scale | 4 months
  Self-rated measurements of social anxiety/phobia.
Change from baseline in Social Phobia Scale + Social Interaction Anxiety Scale | 2 weeks into treatment
  Self-rated measurements of social anxiety/phobia.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | 24 hours
  9-item depression rating scale.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | 11 weeks
  9-item depression rating scale.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | 4 months
  9-item depression rating scale.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | 2 weeks into treatment
  9-item depression rating scale.
Change from baseline in mini-SPIN | Daily, 1-15 days into treatment
  Mini-SPIN is a three-item self-rating scale for assessment of symptoms of social phobia using a five-point Likert scale.
Change from baseline in mini-SPIN | 11 weeks
  Mini-SPIN is a three-item self-rating scale for assessment of symptoms of social phobia using a five-point Likert scale.
Change from baseline in mini-SPIN | 4 months
  Mini-SPIN is a three-item self-rating scale for assessment of symptoms of social phobia using a five-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Per Carlbring, Professor, Principal Investigator — Department of Psychology, Umeå University
Locations (1):
- Department of Psychology, Umeå University, Umeå, Västerbotten County, Sweden

REFERENCES:
- [Background] Boettcher J, Andersson G, Carlbring P; SOFIE-13 Research Group. Combining attention training with cognitive-behavior therapy in Internet-based self-help for social anxiety: study protocol for a randomized controlled trial. Trials. 2013 Mar 8;14:68. doi: 10.1186/1745-6215-14-68. PMID 23497513
- [Result] Boettcher J, Hasselrot J, Sund E, Andersson G, Carlbring P. Combining attention training with internet-based cognitive-behavioural self-help for social anxiety: a randomised controlled trial. Cogn Behav Ther. 2014;43(1):34-48. doi: 10.1080/16506073.2013.809141. Epub 2013 Jul 30. PMID 23898817